CLINICAL TRIAL: NCT04283058
Title: Low Dose Ketamine Infusion for the Treatment of Resistant Depression
Status: Withdrawn | Type: Observational
Why Stopped: Covid-19 disruption of team
Sponsor: Loma Linda University (Other)
Collaborators: Sarah Capalla (Unknown); Ebony HIllery (Unknown); Kaushik Mukherjee (Unknown); Timothy Lee (Unknown)
Responsible Party: Principal Investigator, Patti Radovich, Director of Nursing Research, Loma Linda University
Other Study IDs: LomaLindaU
Record Dates: First submitted 2020-02-21; First posted 2020-02-25 (Actual); Last update posted 2020-05-01 (Actual); Status verified 2020-04

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Ketamine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: Ketamine — d. Ketamine 0.5mg/kg* dose IV in 50 mL NS will be infused at a set non-titratable rate over 40 minutes or Ketamine 1mg/kg* dose IV in 50 mL NS will be infused at a set rate non-titratable over 90 minutes. The dose that the subject will receive will be determined by the Intensive Care Unit Attending based on patient symptoms. Ketamine administered at these doses may result in the following adverse reactions such as excessive sedation or drowsiness, or unpleasant hallucinations, agitation or dysphoric reaction, nausea or increased oral secretions.
  Other Names: Ketalar; Dissaciative anesthetic

SUMMARY:
The purpose of this investigator-initiated observational study is to examine how low Ketamine infusion treatments impact antidepressant and anti-suicidal effects for refractory and non-refractory depression.

DETAILED DESCRIPTION:
This is a descriptive research study that will be collecting prospective outcome data in patients who have been examined Psychiatry and the Intensive Care Unit attending. This study will follow the patients examined and screened by both Psychiatry and the Intensive Care Unit attending physician with orders for the use of ketamine bolus. This study will be examining outcomes of the treatment and will be conducted within adult patients The electronic health records will be reviewed for follow up.

The Primary Objective is to examine the use of Ketamine and the patient outcomes following treatment in individuals with treatment resistant depression. The subjects with treatment resistant depression will be identified by Psychiatric Consult using the Quick Inventory of Depressive Symptomatology evaluation tool, have treatment resistant depression, no history of psychosis, no active substance use, admitted to medical floor and confirmed acceptance to a local Behavioral Medical Center.

Procedures involved (Research Interventions):

Psychiatric consult that includes:

1. A full diagnostic psychiatric interview will be conducted to determine referral appropriateness and discuss other options
2. Review of systems and medical history completed
3. Discussion of treatment alternatives
4. Discussion of off-label use of Ketamine for treatment resistant depression
5. Any necessary labs or additional consults will be suggested at this time. .
6. Review the need to remain NPO for 8 hours prior to treatment and not to take benzodiazepines (i.e., Ativan, Valium, Xanax, Klonopin), alcohol or narcotics (i.e., oxycodone, oxycontin, dilaudid, etc.) within 8 hours of the treatment with the patient.
7. Vitals Assessed on Evaluation - Cardiovascular parameters

   1. Resting systolic BP between 90 and 150
   2. Resting diastolic between 50 and 90 on exam.
   3. If BP is above these parameters, will recommend hypertension be addressed with patient's primary team prior to treatment.

      Quick Inventory of Depressive Symptomology Evaluation (see attached evaluation tool)

      Infusion of Ketamine per physician orders:
   4. Ketamine 0.5mg/kg* dose IV in 50 mL NS will be infused at a set non-titratable rate over 40 minutes or Ketamine 1mg/kg* dose IV in 50 mL NS will be infused at a set rate non-titratable over 90 minutes. The dose that the subject will receive will be determined by the Intensive Care Unit Attending based on patient symptoms. Ketamine administered at these doses may result in the following adverse reactions such as excessive sedation or drowsiness, or unpleasant hallucinations, agitation or dysphoric reaction, nausea or increased oral secretions.

Data collection procedures: The following items will be extracted from the patient's electronic health record: The Quick Inventory of Depressive Symptomatology (QIDS SR-16) completed pre and 24 hours post infusion by Psychiatry MD, vital signs pre, every 15 minutes during infusion and within 5 minutes of completion of infusion and every 15 minutes after until patient is has a PARS of 8 or greater or is back to baseline.

Each subject will be given a unique identification number that will be used on all data collection forms post procedure (infusion). The data will be de- identified after data analysis. The key code will be stored in a separate location from the data stored in secure drive on hospital computer.

Individual subjects may benefit by treatment of their depression. Societal benefits will be an increase in provider knowledge of the effect of this treatment for resistant depression and the ability to quickly treat depression in an acute care setting.

References

1. Kishimoto, T., et al., Single-dose infusion ketamine and non-ketamine N-methyl-d-aspartate receptor antagonists for unipolar and bipolar depression: a meta-analysis of efficacy, safety and time trajectories. Psychological Medicine, 2016. 46(7): p. 1459-1472.
2. Fond, G., et al., Ketamine administration in depressive disorders: a systematic review and meta-analysis. Psychopharmacology (Berl), 2014. 231(18): p. 3663-76.
3. Han, Y., et al., Efficacy of ketamine in the rapid treatment of major depressive disorder: a meta-analysis of randomized, double-blind, placebo-controlled studies. Neuropsychiatr Dis Treat, 2016. 12: p. 2859-2867.
4. Sanacora, G., et al., A Consensus Statement on the Use of Ketamine in the Treatment of Mood Disorders. JAMA Psychiatry, 2017. 74(4): p. 399-405.

ELIGIBILITY:
Inclusion Criteria:

* treatment resistant depression

Exclusion Criteria:

* Patients excluded by SICU/ER attending for treatment based on the following relative contraindications:

  1. Coronary artery disease
  2. Increased intraocular pressure (glaucoma)
  3. Increased intracranial pressure
  4. Uncontrolled hypertension
  5. Kidney dysfunction
  6. Liver dysfunction
  7. Cardiac decompensation
  8. Psychotic disorders (needs further evaluation)

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: treatment resistant depression
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-06-29 (Estimated); Primary Completion 2020-12-29 (Estimated); Study Completion 2020-12-29 (Estimated)

PRIMARY OUTCOMES:
Change in Participants Depressive Symptoms | within 24 hours
  The number of participants treated with Ketamine will have a change in their depressive symptoms using The Quick Inventory of Depressive Symptomatology (QIDS SR-16) completed pre and 24 hours post infusion by Psychiatry MD, vital signs pre, every 15 minutes during infusion and within 5 minutes of completion of infusion and every 15 minutes after until patient is has a PARS of 8 or greater or is back to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Radovich, PhD, Principal Investigator — Loma Linda University Medical Center
Locations (1):
- Loma Linda University Medical Center, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No